CLINICAL TRIAL: NCT02108496
Title: The VENUS Clinical Study (Verifying the Effectiveness of the NUsurface® System) A Multi-centered, Prospective, Randomized, Interventional, Superiority Clinical Study
Brief Title: Verifying the Effectiveness of the NUsurface® System
Acronym: VENUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Active Implants (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000249
Record Dates: First submitted 2014-04-07; First posted 2014-04-09 (Estimated); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Meniscectomy; Osteoarthritis
Keywords: meniscectomy; meniscus; implant; koos; nusurface
MeSH Terms: conditions — Osteoarthritis | interventions — Injections, Intra-Articular; Adrenal Cortex Hormones; Hyaluronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Investigational arm (Experimental): The patients randomized to the Investigational Group will receive the NUsurface® Meniscus Implant.
  Interventions: Device: NUsurface® Meniscus Implant
- Control Arm (Active Comparator): The patients randomized to the Control Group of the study will receive Non-Surgical Care (the current standard of care for this patient population).
  Interventions: Drug: NSAID's and Non-surgical Treatment Options; Drug: Intra-Articular Injections with Corticosteroids; Drug: Intra-Articular Injections with Hyaluronic Acid (HA)

INTERVENTIONS:
Device: NUsurface® Meniscus Implant — The NUsurface Meniscus Implant is a Polycarbonate-Urethane (PCU)-based device reinforced with high tensile Ultra High Molecular Weight Polyethylene (UHMWPE) fibers. The product is available in different sizes, left and right, and with trials so as to allow the surgeon several size options for implantation. The NUsurface® Meniscus Implant, is designed to be conceptually analogous to the natural meniscus whose structural characteristics include a highly orientated collagen fiber network supports the large hoop stresses to produce better distribution of contact pressures within the knee joint. Restoring the distribution of joint loads post-meniscectomy is thought to reducing joint overload and to reducing pain.
  Arms: Investigational arm
Drug: NSAID's and Non-surgical Treatment Options — Non-prescription drugs, creams, vitamins, and supplements, Prescription or Non-Prescriptions NSAIDs, Non-weight bearing and/or open chain physical therapy or self-administered exercise
  Arms: Control Arm
Drug: Intra-Articular Injections with Corticosteroids — Intra-articular injection of a corticosteroid, such as 40 mg of Triamcinolone (e.g. Aristocort or Kenalog).
  Arms: Control Arm
Drug: Intra-Articular Injections with Hyaluronic Acid (HA) — Intra-articular injection of a hyaluronic acid treatment, such as SYNVISC® HA Injections.
  Arms: Control Arm

SUMMARY:
The NUsurface® Meniscus Implant Randomized Study is a multi-center, prospective randomized, interventional clinical trial to test the hypothesis that the NUsurface implant is superior to the non-surgical standard of care in treating the target population.The rationale for performing this clinical study is to gather clinical data to evaluate the safety and effectiveness of the NUsurface device compared to the Standard of Care.

DETAILED DESCRIPTION:
The NUsurface® Meniscus Implant is intended for use in patients with medial compartment pain that have had a previous partial medial meniscectomy.

Patients who meet the inclusion/exclusion criteria will be assigned by balanced randomization into one of two groups: the Meniscus Implants versus non-surgical standard of care. The KOOS (Knee injury and Osteoarthritis Outcome Score) and IKDC (International Knee Documentation Committee) forms will be used to provide a comprehensive evaluation of the patients' pre-intervention and post-intervention condition including activity levels, pain, swelling, locking, stability, support, sports activity, and quality of life assessment.

ELIGIBILITY:
Inclusion Criteria:

* Had > 6 months ago a medial partial meniscectomy as confirmed by patient history and MRI
* Is between age 30 and 75 years (inclusive) at the time of study treatment
* Has neutral alignment ±5º of the mechanical axis, as measured from the angle formed by a line drawn from the center of the femoral head to the medial tibial spine and a line drawn from the medial tibial spine and the center of the ankle joint
* Has ≥ 2 mm intact medial meniscal rim capable of being fitted with a NUsurface® device AND is also recommended for the baseline non-surgical (and, if likely to receive benefit, any injection) therapies to be administered in the study.
* Is willing to be entered into either arm of the study: implanted with the NUsurface device OR treated with the recommended control arm therapies.
* Is willing and able to attend all follow up visits, complete all study questionnaires, and undergo required X-ray and MRI schedule
* Is able and willing to understand and sign the Informed Consent Form
* Is able to read and understand the English language
* Has a KOOS Pain of ≤ 75 (100 being the highest attainable and no pain)

Exclusion Criteria:

* Has a symptomatic knee because of a tear that could be addressed by a repeat partial meniscectomy leaving > 4 mm of medial meniscus rim
* Has evidence of a Outerbridge Grade IV cartilage loss on the medial tibial plateau or femoral condyle that potentially could contact a NUsurface implant (e.g., a focal lesion > 0.5 cm2 correlating to a circular defect of > 8 mm in diameter)
* Has complete disruption of the posterior root attachment of the meniscus
* Has lateral compartment pain and Grade III or Grade IV Outerbridge cartilage score in the lateral compartment
* Has a varus or valgus knee deformity > 5º requiring a tibial or femoral osteotomy
* Has a laxity level of more than Grade II (IKDC), primary or secondary to an injury of the anterior cruciate ligament (ACL) and/or posterior cruciate ligament (PCL) and/or lateral collateral ligament (LCL) and/or medial collateral ligament (MCL)
* Has significant trochlear dysplasia, patellar instability or symptomatic patellar misalignment
* Has patellar compartment pain and Grade III or Grade IV Outerbridge cartilage score in the patellar compartment.
* Compared to a normal knee, has obvious radiological evidence of medial femoral squaring, anatomical variance in the medial tibial plateau, or irregularly shaped cartilage surface
* Had an ACL reconstruction performed < 9 months prior to study treatment
* Has a BMI > 32.5 at the time of study treatment
* Decides to receive (if eligible and an option) allograft medial meniscus transplantation
* Received any type of prosthetic knee implant made of artificial non-resorbable plastic, metal or ceramic, not including the NUsurface® Meniscus Implant
* Has a knee flexion contracture > 10º
* Has flexion < 90º
* Had a previous medial femoral condyle surgery (not including microfracture) or High Tibial Osteotomy (HTO)
* Has insufficiency fractures or avascular necrosis of the medial compartment
* Has an active infection or tumor (local or systemic)
* Has any type of knee joint inflammatory disease including Sjogren's syndrome
* Has neuropathic knee osteoarthropathy, also known as Charcot joint
* Has any medical condition that does not allow possible arthroscopy of the knee
* Has neurological deficit (sensory, motor, or reflex)
* Is currently involved in another investigation of the lower extremity
* Anticipates having another lower extremity surgery during the study period
* Is contraindicated for hyaluronic acid injections (i.e., patients with known hypersensitivity [allergy] to hyaluronan [sodium hyaluronate] preparations); patients having knee joint infections or skin diseases or infections in the site of possible injections
* Is contraindicated for corticosteroid injections (i.e., patients with allergy to any of the components or with idiopathic thrombocytopenic purpura)
* Has received any corticosteroid knee injections ≤ 3 months prior to study treatment
* Has chondrocalcinosis
* Is on immunostimulating or immunosuppressing agents
* Has ipsilateral or contralateral lower limb joint conditions that may affect ambulation or KOOS (e.g. have a leg length discrepancy > 2.5 cm [1 inch], causing a noticeable limp)
* Is a female who is lactating, expecting, or is intending to become pregnant during the study period
* Is an active smoker
* Is mentally incapacitated (incapable of appraising or controlling conduct) or have mental disability (e.g., dementia or Alzheimer's)
* Is a prisoner
* Is a patient who has economic incentive not to improve

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
KOOS Scale | 2 years
  The KOOS Pain Subscale and KOOS Overall Scale (Average of the 5 KOOS Subscales) relative to baseline - all at 24 months.
NUsurface Device Related Complications | 2 years
  The device related complications of the NUsurface Meniscus Implant during the 24-month post-operative period in regard to secondary surgical intervention of the NUsurface device.

CONTACTS AND LOCATIONS:
Overall Officials: Elliott B Hershman, MD, Principal Investigator — Lenox Hill Hospital NYC
Locations (9):
- United States (9):
  - OrthoIndy, Indianapolis, Indiana
  - Brigham and Woman's Hospital, Boston, Massachusetts
  - New England Baptist Hospital, Roxbury Crossing, Massachusetts
  - Capital Region Orthopaedics, Albany, New York
  - Lenox Hill Hospital, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Ohio State University Medical Center, Columbus, Ohio
  - OrthoSouth, Memphis, Tennessee
  - Advanced Orthopaedics, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shemesh M, Asher R, Zylberberg E, Guilak F, Linder-Ganz E, Elsner JJ. Viscoelastic properties of a synthetic meniscus implant. J Mech Behav Biomed Mater. 2014 Jan;29:42-55. doi: 10.1016/j.jmbbm.2013.08.021. Epub 2013 Sep 3. PMID 24055793
- [Background] Zur G, Linder-Ganz E, Elsner JJ, Shani J, Brenner O, Agar G, Hershman EB, Arnoczky SP, Guilak F, Shterling A. Chondroprotective effects of a polycarbonate-urethane meniscal implant: histopathological results in a sheep model. Knee Surg Sports Traumatol Arthrosc. 2011 Feb;19(2):255-63. doi: 10.1007/s00167-010-1210-5. Epub 2010 Jul 16. PMID 20635076
- [Background] Elsner JJ, Portnoy S, Guilak F, Shterling A, Linder-Ganz E. MRI-based characterization of bone anatomy in the human knee for size matching of a medial meniscal implant. J Biomech Eng. 2010 Oct;132(10):101008. doi: 10.1115/1.4002490. PMID 20887018
- [Background] Elsner JJ, Portnoy S, Zur G, Guilak F, Shterling A, Linder-Ganz E. Design of a free-floating polycarbonate-urethane meniscal implant using finite element modeling and experimental validation. J Biomech Eng. 2010 Sep;132(9):095001. doi: 10.1115/1.4001892. PMID 20815651
- [Background] Linder-Ganz E, Elsner JJ, Danino A, Guilak F, Shterling A. A novel quantitative approach for evaluating contact mechanics of meniscal replacements. J Biomech Eng. 2010 Feb;132(2):024501. doi: 10.1115/1.4000407. PMID 20370247
- [Background] Elsner JJ, Shemesh M, Shefy-Peleg A, Gabet Y, Zylberberg E, Linder-Ganz E. Quantification of in vitro wear of a synthetic meniscus implant using gravimetric and micro-CT measurements. J Mech Behav Biomed Mater. 2015 Sep;49:310-20. doi: 10.1016/j.jmbbm.2015.05.017. Epub 2015 May 28. PMID 26057364
- [Result] De Coninck T, Elsner JJ, Linder-Ganz E, Cromheecke M, Shemesh M, Huysse W, Verdonk R, Verstraete K, Verdonk P. In-vivo evaluation of the kinematic behavior of an artificial medial meniscus implant: A pilot study using open-MRI. Clin Biomech (Bristol). 2014 Sep;29(8):898-905. doi: 10.1016/j.clinbiomech.2014.07.001. Epub 2014 Jul 17. PMID 25238685